CLINICAL TRIAL: NCT06511947
Title: An Open-label Phase 1 Trial to Determine the Pharmacokinetics, Pharmacodynamics, and Safety of GH001 Administered Via a Proprietary Aerosol Delivery Device in Healthy Subjects
Brief Title: Pharmacokinetics of GH001 Delivered Via a Proprietary Aerosol Delivery Device in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH001-HV-106-2; IRAS Number (Other: 1009720)
Record Dates: First submitted 2024-06-28; First posted 2024-07-22 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
Keywords: Mebufotenin; 5-MeO-DMT; 5-methoxy-N,N-dimethyltryptamine; GH001; Healthy volunteers; Pharmacokinetics
MeSH Terms: interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Intervention Model Description: This study will include separate single- and multiple-dose parts.
  Part 1 (Single-Dose Part):
  An open-label, non-randomized, parallel design where subjects will be assigned to receive single doses of GH001 delivered via a proprietary aerosol delivery device on a single day in three consecutive cohorts (Cohorts A, B, and C) with eight subjects per cohort. Up to two additional cohorts (Cohorts D and E) may be added before Part 2 is initiated.
  Part 2 (Multiple-Dose Part):
  An open-label, non-randomized design where up to three escalating doses of GH001 will be administered to subjects via a proprietary aerosol delivery device on a single day in one cohort of 12 subjects (Cohort F).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1, Cohort A (Experimental): A single dose inhaled dose of 6 mg GH001 administered via a proprietary aerosol delivery device in eight subjects.
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Part 1, Cohort B (Experimental): A single dose inhaled dose of 12 mg GH001 administered via a proprietary aerosol delivery device in eight subjects.
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Part 1, Cohort C (Experimental): A single dose inhaled dose of 18 mg GH001 administered via a proprietary aerosol delivery device in eight subjects.
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Part 1, Cohort D (optional) (Experimental): A single inhaled intermediate dose of 8, 9, 10, 14, 15, or 16 mg GH001 administered via a proprietary aerosol delivery device in eight subjects (optional cohort dependent on study safety group [SSG] review of PK, PD and safety data from Cohorts A, B, and C).
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Part 1, Cohort E (optional) (Experimental): A single inhaled intermediate dose of 8, 9, 10, 14, 15, or 16 mg GH001 administered via a proprietary aerosol delivery device in eight subjects (optional cohort dependent on SSG review of PK, PD and safety data from Cohorts A, B, and C).
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Part 2, Cohort F (Experimental): Up to three escalating inhaled doses of GH001 (doses as determined by Part 1, maximum single inhaled dose of 18 mg) administered via a proprietary aerosol delivery device in 12 subjects.
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine

INTERVENTIONS:
Drug: 5 Methoxy N,N Dimethyltryptamine — GH001 administered via inhalation
  Other Names: Mebufotenin, 5-MeO-DMT, GH001

SUMMARY:
The primary objectives of this trial are to determine the pharmacokinetic (PK) profile and the safety and tolerability of GH001 delivered via a proprietary aerosol delivery device in healthy subjects after single-dose administration and a single-day individualized dosing regimen (IDR). As secondary objectives, the mebufotenin PK/ pharmacodynamic (PD) relationship, the PD profile of GH001 as evaluated by its psychoactive effects (PsE), the impact on cognitive performance, and the TCmax/2 and TCmax/10 (time taken for Cmax to decrease by 50 and 90%, respectively) are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) in the range of 18.5 to 35 kg/m2 (inclusive) at screening
* Good mental health in the opinion of the investigator.
* Normal spirometry (FEV1 of >80% of predicted and FVC of >80% of predicted value) at screening.

Exclusion Criteria:

* Has known allergies or hypersensitivity or any other contraindication to mebufotenin, bufotenin, melatonin or triptans.
* Has received any investigational medication, including investigational vaccines, in the 3 months prior to baseline or is in the follow-up period of another clinical trial at the time of screening for this trial.
* Has a current or past clinically significant condition, which renders the subject unsuitable for the trial according to the investigator's judgement.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Serum PK parameters of mebufotenin - maximum observed concentration (Cmax) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - time of maximum observed concentration (Tmax) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - terminal elimination half-life (t1/2) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - area under the serum concentration-time curve from time zero to the last quantifiable concentration (AUC0-t) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - area under the serum concentration-time curve extrapolated to infinity (AUC0-∞) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - terminal elimination rate constant (λz) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - apparent total body clearance (CL/F) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - apparent steady-state volume of distribution (VSS/F) | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Serum PK parameters of mebufotenin - Cmax/AUC0-∞ | Up to 6 hours
  For PK analyses, blood samples will be collected before and up to 6 hours after the administration of GH001 to determine mebufotenin serum concentrations.
Safety and tolerability: incidence of treatment-emergent adverse events | Up to 7 days
  Adverse events reported in the study and coded by MedDRA.
Safety and tolerability: clinically significant changes from baseline in electrocardiogram (ECG), vital signs, spirometry and safety laboratory assessments | Up to 7 days
  Percentage of subjects with clinically significant changes* from baseline in ECG (heart rate, RR, QT, PR, and QRS intervals, and QTcF).
  Percentage of subjects with clinically significant changes* from baseline in vital signs (systolic and diastolic blood pressure, respiration rate, heart rate, peripheral oxygen saturation, body temperature).
  Percentage of subjects with clinically significant changes* from baseline in spirometry (forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC]).
  Percentage of subjects with clinically significant changes* from baseline in safety laboratory assessments (hematology, biochemistry, and urinalysis).
  *Clinically significant changes as determined by the principal investigator
Safety and tolerability: assessment of sedation (Modified Observer's Assessment of Alertness and Sedation [MOAA/S]) following each dose and as part of the discharge evaluation on Day 0 | Postdose, up to discharge on dosing day (Day 0)
  The MOAA/S will be completed before and after GH001 dosing. Scored from 0 (deep sedation) to 5 (alert).
Safety and tolerability: change from baseline in Clinician Administered Dissociative States Scale (CADSS) | From baseline up to 7 days
  The CADSS comprises 19 subjective items, ranging from 0 'not at all' to 4 'extremely. Summed together, these subscales form a total dissociative score. Combined score ranges from 0 to 76.
Safety and tolerability: assessment of subject discharge readiness at discharge on Day 0 | Postdose, at discharge on dosing day (Day 0)
  Assessment of Discharge Readiness on the administration day by the principal investigator, using the Clinical Assessment of Discharge Readiness (CADR).
Safety and tolerability: Columbia-Suicide Severity Rating Scale (C-SSRS) categorization. | Up to 7 days
  A detailed questionnaire assessing both suicidal behaviour and suicidal ideation.
Safety and tolerability: Change from baseline in Brief Psychiatric Rating Scale (BPRS). | From baseline up to 7 days
  A scale to measure psychiatric symptoms. Each symptom is rated 1-7 and a total of 18 symptoms are scored. Combined score ranges from 18 to 126 and a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- GH Research Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No